CLINICAL TRIAL: NCT06261645
Title: ROTOFUNC - a Randomized and Controlled Study to Evaluate the Effect of a Novel Assessment and Treatment Strategy for Patients With Non-traumatic Shoulder Instability
Brief Title: Rotofunc - Non-traumatic Shoulder Instability and Total Rotator Cuff Function
Acronym: ROTOFUNC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Ingrid Hultenheim Klintberg, Principal Investigator, Sahlgrenska University Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ROTOFUNK_2_2023
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Shoulder Dislocation or Subluxation
Keywords: physiotherapy; muscle control; non-surgical
MeSH Terms: conditions — Shoulder Dislocation; Joint Dislocations

STUDY DESIGN:
Intervention Model Description: A 16 week exercise program with specific exercises to restore total rotator cuff function individually selected during clinical physiotherapy visits and performed 2 - 4 times daily.
  In addition, the patient will receive education and guidance in the daily use of the arm to adjust to appropriate load on the shoulder.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator: 6 physiotherapists are care providers, responsible for the Intervention . Two independent investigators does not know who is the actual care provider. However, all patients recieve the same intervention.
  Outcome assessor: each participant is given a research code. The results from the assessments are entered in the data base by a research assistant, not involved in the study on any level.
  Individuals are not identifiable. The outcome assessor are planning for all statistics used and is not in other ways involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early start (Experimental): According to result from the random allocation patients in Early Start will initiate their treatment within two weeks following the Baseline assessment.The intervention consists of a 16 week exercise program with specific exercises to restore total rotator cuff function individually selected during clinical physiotherapy visits and performed 2 - 4 times daily.
  According to progression, a mean of 10 visits are anticipated over the 16 weeks In addition, the patient will receive education and guidance in the daily use of the arm to adjust to appropriate load on the shoulder.
  Interventions: Other: Early Physiotherapist selected active exercises
- Delayed start (Experimental): According to result from the random allocation patients in Delayed Start will delay the start of their treatment with 16 weeks.
  Participants in Delayed Start will undergo the same Baseline assessment a second time, and initiate their treatment within 2 weeks thereafter. The intervention consists of a 16 week exercise program with specific exercises to restore total rotator cuff function individually selected during clinical physiotherapy visits and performed 2 - 4 times daily.
  According to progression, a mean of 10 visits are anticipated over the 16 weeks In addition, the patient will receive education and guidance in the daily use of the arm to adjust to appropriate load on the shoulder.
  Interventions: Other: Delayed Physiotherapist selected active exercises

INTERVENTIONS:
Other: Early Physiotherapist selected active exercises — Exercises to restore total rotator cuff function selected and progressed according to patients performance. Performance is assessed by the physiotherapist regarding available range of motion, comfort during as well as pain-free performance.
  Education on shoulder muscles functional anatomy and on effect of pain on muscle performance
  Arms: Early start
Other: Delayed Physiotherapist selected active exercises — Exercises to restore total rotator cuff function selected and progressed according to patients performance. Performance is assessed by the physiotherapist regarding available range of motion, comfort during as well as pain-free performance.
  Education on shoulder muscles functional anatomy and on effect of pain on muscle performance
  Arms: Delayed start

SUMMARY:
The goal of this clinical trial is to test the effect of a novel assessment and treatment strategy for young adults with severely disabling non-traumatic shoulder instability. The main question it aims to answer is if this treatment will substantially change the patients shoulder function to a more stable and controllable state and thereby give a higher quality of life. Participants failure in active shoulder muscle function will be assessed and exercises will be selected individually. Patients will be asked to perform the exercises twice per day. At clinical visits to a specialized physiotherapist the exercises will be upgraded to restore full dynamic stability throughout shoulder movement range. The active treatment period will be 4 months. Researchers will compare two groups. One group will start directly after a baseline assessment is fulfilled. The other group will receive the treatment with a delay of 4 months to evaluate if the selected exercises can substantially change the shoulder stability compared to no treatment, the natural course of the condition.

DETAILED DESCRIPTION:
Impaired shoulder function and pain results in decreased quality-of-life, reduced working capacity and affect both society and individuals with high costs. Young adults with non-traumatic shoulder instability are one of the most difficult patient groups to treat. Surgery has previously been the treatment offered for these patients. Today, surgery is more and more questioned and physiotherapy and now active exercises are suggested to be the first - line of treatment.

A novel physiotherapy treatment strategy has been developed during the recent years.

The intervention is based on an entirely updated mode to assess and restore shoulder muscle function. The development has been initiated by new data from EMG- studies that has given a deepened understanding of the complex stabilizing muscle function of the shoulder. The hypothesis is that the main stabilizing muscles, the rotator cuff has by franc dislocations, subluxations and pain lost its rapidness, precision, and endurance to keep the humeral head stabilized and centered within the glenoid fossa.

The hypothesis is that with restored, full rotator cuff function, i. e. a rotator cuff able to perform its stabilizing role and the mover role into the extremes of the range of motion, where the fibers act from their most shortened to their most lengthened positions and during concentric as well as eccentric muscle action, will regain the sense of shoulder stability, pain-free shoulder function and higher quality-of-life.

The purpose of this study is to evaluate the effect of this new active exercise-based intervention in patients with non-traumatic shoulder instability.

Methods: A total of 100 patients randomly be allocated into two different groups, Early start and Delayed start. Both groups will receive the same 16-week physiotherapy supervised exercise program, however the latter group with a delay of four months.

The primary outcome is assessment of neuromuscular control during active rotation movements documented with video. The range of motion is measured, and sway and steadiness are graded. The secondary outcomes include: 1) active and passive range of motion; 2) shoulder pain at rest using an 11-graded numeric rating scale; 3) Pain during motion, and 4) Apprehension during motion using Patient Specific Functional Scale; 5) Quality-of-life will be assessed using Western Ontario Shoulder Instability Index (WOSI) Patients will be assessed by one of two independent investigators at baseline (second baseline if Delayed Start), 6 weeks, 4 and 12 months. At 4 and 12 months also Patient's Satisfaction of being treated with the novel strategy will be assessed.

The statistical analysis will assess change over time and differences between groups using ANOVA and Tukey's PostHoc-test as well as Kruskal- Wallis and Mann-Whitney-U test with the significant level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* young adults, non traumatic as well as non-controllable, positional, functional shoulder instability according to Moroder et al. demonstrating a lack of ≥ 20%, active, dynamic control compared with the total passive range of motion in shoulder rotation with or without previous shoulder stabilizing surgery
* Understanding the Swedish language well, in speaking, in reading and writing.

Exclusion Criteria:

* Other significant shoulder pathologies, patients diagnosed with severe systemic connective tissue, congenital anatomic abnormalities, or psychiatric diagnoses according to previous medical records
* <60% adherence to assigned exercises

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular control | Baseline One, Baseline Two (Delayed start,DS), 4 and 12 months
  Available range of motion during shoulder rotation during 8 different test situations, in prone and in supine with support and without support for the upper arm (degrees). The performance, sway and halting during motion, will be graded using a Likert scale: no deviation, small deviation, medium- or important deviation from optimal non-symptomatic shoulder function.

SECONDARY OUTCOMES:
Clinical assessment - Active and passive range of motion | Baseline One, Baseline Two (DS), 4 and 12 months
  will be assessed in standing and in lying supine in both shoulders. Flexion, abduction and external and internal rotation with shoulders at 90° abduction.
Pain at rest | Baseline One, Baseline Two (DS) 6 weeks, 4 and 12 months
  - during the last week will be assessed using an 11-graded numeric rating scale (NRS).
Pain during motion | Baseline One, Baseline Two (DS) 6 weeks, 4 and 12 months
  Four activities that affect the patients every-day life will be selected and assessed using Patient Specific Functional scale, each graded 0 -10, with a higher score indicating higher, better function.
Apprehension of instability during motion | Baseline One, Baseline Two (DS) 6 weeks, 4 and 12 months
  Four activities that affects the patients every-day life by discomfort and apprehension will be selected and assessed using Patient Specific Functional scale, each graded 0 -10, with a higher score indicating higher, better function.
Patient reported quality-of-life in relation to shoulder function | Baseline One, Baseline Two (DS) 6 weeks, 4 and 12 months
  - will be assessed using Western Ontario Shoulder Instability Index [9]. The questionnaire consists of 21 items. Patients rate their percieved function for each item using Visual Analogue Scales, 0 - 100 mm, with a lower score indicating better function. The result of the total score is presented in percentage of full (100%) shoulder function i.e. perceived quality of life using related to shoulder function. Higher percent indicates better function.
Patient's satisfaction | At 4 and 12 months
  - of being treated according to the novel concept will be assessed using a five-graded Likert scale: Very dissatisfied; Dissatisfied; neither dissatisfied nor satisfied; Satisfied and Very satisfied.
  As well as: Would you recommend this treatment concept to a friend or relative with similar shoulder dysfunction as yours?, will be assessed using the three response options: Yes, No, or Do not know

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fagevik Olsén, Professor, Principal Investigator — Sahlgrenska Academy, Inst Neuroscience and Physiology/Physiotherapy
Locations (1):
- Sahlgrenska University Hospital/Mölndal, Physiotherapy Dpt, Gothenburg, Mölndal, Sweden

REFERENCES:
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Result] Boettcher CE, Ginn KA, Cathers I. Which is the optimal exercise to strengthen supraspinatus? Med Sci Sports Exerc. 2009 Nov;41(11):1979-83. doi: 10.1249/MSS.0b013e3181a740a7. PMID 19812522
- [Result] Moroder P, Danzinger V, Maziak N, Plachel F, Pauly S, Scheibel M, Minkus M. Characteristics of functional shoulder instability. J Shoulder Elbow Surg. 2020 Jan;29(1):68-78. doi: 10.1016/j.jse.2019.05.025. Epub 2019 Aug 1. PMID 31378683
- [Result] Boettcher CE, Cathers I, Ginn KA. The role of shoulder muscles is task specific. J Sci Med Sport. 2010 Nov;13(6):651-6. doi: 10.1016/j.jsams.2010.03.008. Epub 2010 May 7. PMID 20452282
- [Result] Dark A, Ginn KA, Halaki M. Shoulder muscle recruitment patterns during commonly used rotator cuff exercises: an electromyographic study. Phys Ther. 2007 Aug;87(8):1039-46. doi: 10.2522/ptj.20060068. Epub 2007 Jun 19. PMID 17578940
- [Result] Dube JA, Mercier C. Effect of pain and pain expectation on primary motor cortex excitability. Clin Neurophysiol. 2011 Nov;122(11):2318-23. doi: 10.1016/j.clinph.2011.03.026. Epub 2011 May 20. PMID 21601513
- [Result] Jaggi A, Herbert RD, Alexander S, Majed A, Butt D, Higgs D, Rudge W, Ginn KA. Arthroscopic capsular shift surgery in patients with atraumatic shoulder joint instability: a randomised, placebo-controlled trial. Br J Sports Med. 2023 Dec;57(23):1484-1489. doi: 10.1136/bjsports-2022-106596. Epub 2023 Jun 12. PMID 37308285
- [Result] Ginn KA, Cathers I, Boettcher C, Halaki M. Analysis of phase detects altered timing of muscle activation in subjects with chronic shoulder pain. J Electromyogr Kinesiol. 2022 Feb;62:102621. doi: 10.1016/j.jelekin.2021.102621. Epub 2021 Nov 22. PMID 34847442
- [Result] Gajdosik RL, Bohannon RW. Clinical measurement of range of motion. Review of goniometry emphasizing reliability and validity. Phys Ther. 1987 Dec;67(12):1867-72. doi: 10.1093/ptj/67.12.1867. PMID 3685114
- [Result] Kirkley A, Griffin S, McLintock H, Ng L. The development and evaluation of a disease-specific quality of life measurement tool for shoulder instability. The Western Ontario Shoulder Instability Index (WOSI). Am J Sports Med. 1998 Nov-Dec;26(6):764-72. doi: 10.1177/03635465980260060501. PMID 9850776
- [Result] Nazari G, Bobos P, Lu Z, Reischl S, MacDermid JC. Psychometric properties of Patient-Specific Functional Scale in patients with upper extremity disorders. A systematic review. Disabil Rehabil. 2022 Jun;44(13):2958-2967. doi: 10.1080/09638288.2020.1851784. Epub 2020 Dec 8. PMID 33290102
- [Result] Wattanaprakornkul D, Halaki M, Cathers I, Ginn KA. Direction-specific recruitment of rotator cuff muscles during bench press and row. J Electromyogr Kinesiol. 2011 Dec;21(6):1041-9. doi: 10.1016/j.jelekin.2011.09.002. Epub 2011 Oct 5. PMID 21978788
- [Result] Wattanaprakornkul D, Cathers I, Halaki M, Ginn KA. The rotator cuff muscles have a direction specific recruitment pattern during shoulder flexion and extension exercises. J Sci Med Sport. 2011 Sep;14(5):376-82. doi: 10.1016/j.jsams.2011.01.001. Epub 2011 Feb 17. PMID 21333595